CLINICAL TRIAL: NCT05268094
Title: Comparison of Methods of Pulmonary Blood Flow Augmentation in Neonates: Shunt Versus Stent (The COMPASS Trial)
Acronym: COMPASS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: Pediatric Heart Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHNCOMPASS
Record Dates: First submitted 2022-01-19; First posted 2022-03-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Congenital Heart Disease in Children
Keywords: Congenital Heart Disease; Ductal Dependent Pulmonary Blood Flow; Ductal Artery Shunt; Systemic-to-Pulmonary Artery Shunt
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either an SPS or DAS. Overall randomization will be 1:1 to each treatment arm, with block randomization will be performed by center and by single vs. two ventricle status
Masking Description: Study staff and participants' families will be aware of treatment group due to the nature of the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Ductal Artery Stent (Experimental): Transcatheter ductal artery shunt will be placed by the interventional team. Drug-eluting coronary stent brand, length, and diameter are determined by the interventional team.
  Interventions: Device: Ductal Arterial Stent
- Systemic-to-Pulmonary Artery Shunt (Experimental): Surgical systemic-to-pulmonary artery shunt performed by the interventional team. SPS diameter, length, and material will be determined by the surgeon performing the intervention.
  Interventions: Procedure: Systemic-to-Pulmonary Artery Shunt

INTERVENTIONS:
Device: Ductal Arterial Stent — Drug-eluting ductal arterial stents will be placed by transcatheter method.
  Other Names: Medtronic Resolute Onyx; Boston Scientific Promus Elite/Premier; Boston Scientific Synergy; Cordis Elunir; Abbott Xience
  Arms: Ductal Artery Stent
Procedure: Systemic-to-Pulmonary Artery Shunt — A surgical connection will be made between a systemic artery and the pulmonary artery.
  Arms: Systemic-to-Pulmonary Artery Shunt

SUMMARY:
COMPASS is a prospective multicenter randomized interventional trial. Participants with ductal-dependent pulmonary blood flow will be randomized to receive either a systemic-to-pulmonary artery shunt or ductal artery stent. Block randomization will be performed by center and by single vs. two ventricle status. Participants will be followed through the first year of life.

DETAILED DESCRIPTION:
In neonates with ductal-dependent blood flow there remains valid uncertainty regarding the comparative benefits of ductal artery stent (DAS) with the traditional systemic-to-pulmonary artery shunt (SPS) palliation due to the lack of previous multicenter studies. COMPASS is a prospective multicenter randomized interventional trial where participants will be randomized to receive either an SPS or DAS to compare rates of a composite major morbidity/mortality endpoint in the first year of life. The study objectives are to perform an intention-to-treat analysis of participants' outcomes, and to describe the failure rate for neonatal candidates for DAS and the impact of this failure on the post-SPS course. Participants will be followed through the first year of life.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates with Congenital Heart Disease (CHD) and ductal-dependent pulmonary blood flow requiring only a stable source of pulmonary blood flow as the initial palliation, for whom the clinical decision is made at the enrolling center that this is best achieved by either DAS or SPS.
2. Age ≤ 30 days at time of index procedure (DAS or SPS).

Exclusion Criteria:

* 1. Any patient for whom the clinical decision at the enrolling center is that an initial intervention other than DAS or SPS is indicated (e.g., Right Ventricle-Pulmonary Artery (RV-PA) conduit, Right Ventricular Outflow Tract (RVOT) stent, primary complete anatomic repair, etc.).

  2. Pulmonary Atresia with Intact Ventricular Septum (PA/IVS) where Right Ventricle (RV) decompression is planned.

  3. Presence of MAPCAs: defined as an aortopulmonary collateral that is expected to require unifocalization.

  4. Non-confluent Pulmonary Arteries (i.e., isolated Pulmonary Artery (PA) of ductal origin).

  5. Acutely jeopardized branch Pulmonary Arteries (>75% narrowing of proximal PA based on screening cross sectional imaging [Computed Tomography Angiography (CTA) or cardiovascular Magnetic Resonance (cMR)]).

  6. Bilateral Patent Ductus Arteriosis (PDA). 7. Patient who, at the time of enrollment, is deemed not to be a candidate for eventual Glenn or Complete Surgical Repair (CSR) for any reason.

  8. Birth weight <2.0 kg. 9. Gestational age <34 weeks at birth. 10. Patient for whom additional intervention is expected concomitant with, or prior to, DAS or SPS (e.g., atrial septostomy, aortic arch intervention, or RV outflow tract intervention) - except for branch PA arterioplasty or stent/balloon angioplasty.

  11. Major co-morbidities which, in the opinion of the investigator, would negatively alter expected 1-year survival (e.g., intracranial hemorrhage, renal failure, etc.).

  12. Specific known genetic anomaly which, in the opinion of the investigator, would be expected to significantly alter clinical course in the first year of life (e.g., Trisomy 13/18, CHARGE, VACTERL).

  13. Patient who does not plan to return to the enrolling center or another participating center for Glenn/CSR.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Morbidity and/or Mortality Endpoint | 1 year
  Rates of a composite major morbidity and/or mortality endpoint in the first year of life will be compared between neonates with ductal-dependent pulmonary blood flow randomized to receive either DAS or SPS as the initial palliation.

SECONDARY OUTCOMES:
Global Rank Score | 1 year
  All participants will be assigned a Global Rank Score, which is a rank based on a pre-specified hierarchical ranking of outcomes. This combines various endpoints into a single quantifiable endpoint with weighting of the severity of the component endpoints, and allows for the inclusion of endpoints of different forms. Global rank scores will range from 1-7.
Freedom from Adverse Events | 1 year
  Safety, defined as freedom from procedural adverse events and complications, will be tracked and evaluated.
Days Alive out of Hospital | 1 year
  Days alive out of the hospital represents a patient-centered outcome, and functions as a composite endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Petit, MD, Study Chair — Columbia University; Andrew Glatz, MD, Study Chair — Washington University School of Medicine; Sara Pasquali, MD, Study Chair — University of Michigan; Jenna Romano, MD, Study Chair — University of Michigan; Jeffrey Zampi, MD, Study Chair — University of Michigan
Locations (24):
- United States (23):
  - University of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospitals, Oakland, California
  - Stanford Children's Health, Palo Alto, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - New York Presbyterian Hospital/Columbia University Irving Medical Center, New York, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadephia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Wisconsin, Wauwatosa, Wisconsin
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected by the Data Coordinating Center will be shared after posting of results and main study results publication.
Supporting Information: Study Protocol, ICF
Time Frame: Protocol and Informed Consent Form will be shared within 12 months of publication of study results. Public Use Dataset will be made available after publication, timeframe to be decided.
Access Criteria: Protocol and Informed Consent Form will be made available with results on clinicaltrials.gov. Public Use Dataset will be available on the Pediatric Heart Network public website and may be used in accordance with Pediatric Heart Network governance.
URL: https://www.pediatricheartnetwork.org/login/

REFERENCES:
- [Derived] Reddy D, Kleinloog R, Kinsley R. Pulmonary Atresia, Ventricular Septal Defect, and Major Aortopulmonary Collateral Arteries: The Natural History and Late Presentation. World J Pediatr Congenit Heart Surg. 2025 Mar;16(2):203-207. doi: 10.1177/21501351241311882. Epub 2025 Feb 4. PMID 39905870
- [Derived] Petit CJ, Romano JC, Zampi JD, Pasquali SK, McCracken CE, Chanani NK, Les AS, Burns KM, Crosby-Thompson A, Stylianou M, Kato B, Glatz AC; Pediatric Heart Network Investigators. Rationale and design of the randomized COmparison of Methods for Pulmonary blood flow Augmentation: Shunt versus Stent (COMPASS) trial: A Pediatric Heart Network study. Catheter Cardiovasc Interv. 2024 Oct;104(4):637-647. doi: 10.1002/ccd.31109. Epub 2024 Sep 23. PMID 39311092
- [Derived] Petit CJ, Romano JC, Zampi JD, Pasquali SK, McCracken CE, Chanani NK, Les AS, Burns KM, Crosby-Thompson A, Stylianou M, Kato B, Glatz AC; Pediatric Heart Network Investigators. Rationale and Design of the Randomized COmparison of Methods for Pulmonary Blood Flow Augmentation: Shunt Versus Stent (COMPASS) Trial: A Pediatric Heart Network Study. World J Pediatr Congenit Heart Surg. 2024 Nov;15(6):693-702. doi: 10.1177/21501351241266110. Epub 2024 Sep 23. PMID 39308140
- See also: Pediatric Heart Network Current Studies — https://www.pediatricheartnetwork.org/studies/